CLINICAL TRIAL: NCT05314855
Title: Role of the Central Brain Clock in the Pathophysiology of Insulin Resistance
Brief Title: Brain Clock and Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dirk Jan Stenvers, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL79698.018.21
Record Dates: First submitted 2022-03-07; First posted 2022-04-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Insulin Resistance; Type 2 Diabetes
Keywords: Type 2 Diabetes Mellitus; Insulin resistance; Suprachiasmatic nucleus; functional MRI
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese individuals with normal insulin sensitivity
  Interventions: Device: functional MRI
- Obese individuals with impaired insulin sensitivity
  Interventions: Device: functional MRI
- Obese patients with type 2 diabetes
  Interventions: Device: functional MRI

INTERVENTIONS:
Device: functional MRI — Subjects will undergo functional MRI at 4 time points in 24 hours.

SUMMARY:
In this observational cohort study the investigators will determine the activity rhythm of the suprachiasmatic nucleus in humans with progressive stages of insulin resistance, using advanced functional brain imaging (7 Tesla functional MRI).

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) has an increasing worldwide incidence. Insulin resistance is a key pathophysiological process in the development of hyperglycemia in patients with T2DM. Disruption of circadian synchrony leads to insulin resistance. Animal studies and post-mortem human brain studies suggest that the master brain clock in the hypothalamic suprachiasmatic nucleus (SCN) plays a role in the development of insulin resistance. Up to now, no-one has investigated whether the in vivo activity rhythm of the SCN is affected in patients with insulin resistance. The investigators hypothesize that the master brain clock has an important role in the development of human insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

Group 1: obese people with normal insulin sensitivity

* age 25-65 years
* BMI>30
* fasting plasma insulin ≤62 pmol/L
* fasting plasma glucose <5.6 mmol/L
* Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) ≤ 4.5

Group 2: obese people with insulin resistance

* age 25-65 years
* BMI>30
* fasting plasma insulin >62 pmol/L
* not fulfilling the American Diabetes Association (ADA) criteria for type 2 DM

Group 3: obese subjects with overt type 2 DM

* age 25-65 years
* BMI>30
* diagnosis type 2 DM according to ADA criteria

Exclusion Criteria:

* An extreme chronotype (midpoint of sleep on free days (MSFsc) before 2:00 or after 6:00).
* Active psychiatric disorder (including circadian rhythm sleep disorder) as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM) 5
* Disorders of the central nervous system (Early-onset dementia, stroke, epilepsy, Parkinson's disease, brain tumor)
* Severe visual impairment (WHO classification)
* Shift workers
* Crossing > 2 time zones in the 3 months before the study
* Patients with type 2 DM receiving insulin treatment or glucagon-like peptide (GLP) 1 agonists
* MRI contraindications

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinics, community sample
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
SCN blood oxygen level dependent (BOLD) response to light: mean SCN activity | mean activity over 24 hours
  SCN BOLD response to light stimulus (percent BOLD signal change)
SCN BOLD response to light: time point of peak SCN activity | 24 hours
  time point (zeitgeber time in hh:mm)
SCN BOLD) response to light: time point of trough SCN activity | 24 hours
  time point (zeitgeber time in hh:mm)
Amplitude of SCN activity rhythm (peak-trough change in SCN activity) | 24 hours
  Peak-trough difference in SCN activity (percent BOLD signal change)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. D.J. Stenvers, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam University Medical Centers, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] World Health Organization, Global report on diabetes., in WHO Library. 2016
- [Background] Cleland SJ, Fisher BM, Colhoun HM, Sattar N, Petrie JR. Insulin resistance in type 1 diabetes: what is 'double diabetes' and what are the risks? Diabetologia. 2013 Jul;56(7):1462-70. doi: 10.1007/s00125-013-2904-2. Epub 2013 Apr 24. PMID 23613085
- [Background] Stenvers DJ, Scheer FAJL, Schrauwen P, la Fleur SE, Kalsbeek A. Circadian clocks and insulin resistance. Nat Rev Endocrinol. 2019 Feb;15(2):75-89. doi: 10.1038/s41574-018-0122-1. PMID 30531917
- [Background] Hogenboom R, Kalsbeek MJ, Korpel NL, de Goede P, Koenen M, Buijs RM, Romijn JA, Swaab DF, Kalsbeek A, Yi CX. Loss of arginine vasopressin- and vasoactive intestinal polypeptide-containing neurons and glial cells in the suprachiasmatic nucleus of individuals with type 2 diabetes. Diabetologia. 2019 Nov;62(11):2088-2093. doi: 10.1007/s00125-019-4953-7. Epub 2019 Jul 20. PMID 31327049
- [Background] ter Horst KW, Gilijamse PW, Koopman KE, de Weijer BA, Brands M, Kootte RS, Romijn JA, Ackermans MT, Nieuwdorp M, Soeters MR, Serlie MJ. Insulin resistance in obesity can be reliably identified from fasting plasma insulin. Int J Obes (Lond). 2015 Dec;39(12):1703-9. doi: 10.1038/ijo.2015.125. Epub 2015 Jul 9. PMID 26155920
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Roenneberg T, Kuehnle T, Pramstaller PP, Ricken J, Havel M, Guth A, Merrow M. A marker for the end of adolescence. Curr Biol. 2004 Dec 29;14(24):R1038-9. doi: 10.1016/j.cub.2004.11.039. No abstract available. PMID 15620633
- [Background] World report on vision. Geneva: World Health Organization. 2019